CLINICAL TRIAL: NCT00011934
Title: Granulocyte-Macrophage Colony Stimulating Factor (Rhu-GM-CSF) and Autologous Bone Marrow Transplantation for Chronic Myeloid Leukemia
Brief Title: Bone Marrow Transplantation Plus Biological Therapy in Treating Patients With Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068460, J9833; P30CA006973 (NIH); JHOC-J9833; IMMUNEX-001.0683; JHOC-98051405; NCI-G01-1912
Record Dates: First submitted 2001-03-03; First posted 2004-05-04 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; sargramostim

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: sargramostim
Procedure: autologous bone marrow transplantation

SUMMARY:
RATIONALE: Biological therapy may increase the number of immune cells found in bone marrow and may help a person's immune system recover from the side effects of the chemotherapy used in treating chronic myeloid leukemia. Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of bone marrow transplantation, chemotherapy, and biological therapy in treating patients who have chronic myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the one year event-free survival in patients with chronic phase chronic myeloid leukemia receiving sargramostim (GM-CSF)-treated autologous bone marrow transplantation followed by GM-CSF and interferon alfa. II. Determine the toxicity of this regimen in these patients.

OUTLINE: Patients undergo harvesting of autologous bone marrow. A portion of the cells are treated ex vivo with sargramostim (GM-CSF) for 3 days. Patients then receive myeloablative chemotherapy with busulfan and cyclophosphamide on days -9 to -2 according to the preparative regimen protocol. Patients undergo sargramostim (GM-CSF)-treated autologous bone marrow transplantation on day 0. Patients receive GM-CSF subcutaneously daily on days 5-180, and interferon alfa daily on days 90-180. Patients are followed monthly for 1 year, every 6 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 9-19 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of chronic phase chronic myeloid leukemia (CML) by cytogenetic and/or molecular analyses No more than 10% blasts on blood and bone marrow morphology Philadelphia (Ph) chromosome positive Ph chromosome-negative CML allowed if evidence of the BCR-ABL rearrangement by molecular or FISH analyses or evidence of the P120 protein Duration of CML less than 3 years, unless cytogenetic remission to interferon has been achieved Failed to obtain and maintain a complete cytogenetic remission on a prior trial of interferon therapy Absence of detectable PH-negative cells in bone marrow or blood after 6 months of therapy Lack of a progressive increase in Ph-negative cells between 6 and 12 months of therapy Less than 50% Ph-negative cells after 12 months of therapy Absence of complete cytogenetic remission after 24 months of therapy Inability to tolerate prior interferon therapy No accelerated phase or blast crisis CML, chronic myelomonocytic leukemia, or juvenile CML Concurrent enrollment on the busulfan and cyclophosphamide preparative regimen protocol

PATIENT CHARACTERISTICS: Age: 12 to 70 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No history of intolerance to sargramostim (GM-CSF)

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-05; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States